CLINICAL TRIAL: NCT04873791
Title: Comparison of Cognitive Function, Balance, Quality of Life, Depression and Daily Living Activities of Geriatric Individuals Living in Home Environment and Nursing Home.
Brief Title: Comparison of the Effects of Different Living Environments in Geriatric Individuals: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 10156977
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Aging Problems; Balance; Distorted; Pain; Quality of Life
Keywords: Geriatric individuals; Nursing home; Home environment; Balance; Pain; Quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Assessment Geriatric Individuals Living at Home were joined in Group 1.
  Demographic and social characteristics, cognitive functions, balance, pain, depression, quality of life, and activities of daily living of elderly individuals living in a nursing home and home environment were evaluated.
  Demographic information of all subjects (age, gender, educational status, occupation, body weight, height, body mass index), Standardized Mini-Mental Test (SMMT) score, Visual Analog Scale (VAS) score, Berg Balance Scale (BBS) score, Geriatric Depression Scale (GDS) score, Barthel Index score, Short Form-36 (SF-36) score were used for evaluations.
  Assessments were made as described in section of outcome measures, in one session.
  Interventions: Diagnostic Test: Assessment of geriatric individuals living in home environment and nursing home.
- Group 2: Assessment Geriatric Individuals Living in Nursing Home were joined in Group 2. Demographic and social characteristics, cognitive functions, balance, pain, depression, quality of life, and activities of daily living of elderly individuals living in a nursing home and home environment were evaluated.
  Demographic information of all subjects (age, gender, educational status, occupation, body weight, height, body mass index), Standardized Mini-Mental Test (SMMT) score, Visual Analog Scale (VAS) score, Berg Balance Scale (BBS) score, Geriatric Depression Scale (GDS) score, Barthel Index score, Short Form-36 (SF-36) score were used for evaluations.
  Assessments were made as described in section of outcome measures, in one session.
  Interventions: Diagnostic Test: Assessment of geriatric individuals living in home environment and nursing home.

INTERVENTIONS:
Diagnostic Test: Assessment of geriatric individuals living in home environment and nursing home. — Assessments explained in the arm section were made as described in one session in both group

SUMMARY:
In Turkey, 63% of geriatric people who make up approximately 8.3% of the entire population live in their own living environment, 36% live with their children and 1% live in nursing homes. The number of individuals living in nursing homes is increasing as the nuclear family structure becomes more evident. National Social Security programs give special importance to nursing home restructuring and Social Health Policy aims to increase practices related to "aging in place" and "Active and Healthy Ageing" for geriatric individuals. In this context, projects aimed at preventing secondary negative symptoms in aging and supporting the quality aging process are outstanding.

The aim of this study is to assess and compare cognitive functions, balance, musculoskeletal pain severity, psychological state, participation level in activities of daily living, and quality of life of geriatric individuals living different environments.

DETAILED DESCRIPTION:
Aging is a process that negatively affects the individual physiologically, psychologically, and socially. Degenerative changes in the musculoskeletal system cause joint pain, limitations, restrictions on activity participation, and physical and social dependence. Neurodegenerative processes, on the other hand, lead to loss of cognitive functions, balance, and coordination. The decrease in biological and social motives and the gradual increase in social and physiological losses, lead to dependence in the activities of daily living, worsening psychological condition, and deteriorating quality of life. With this process, the caregiver burden increases economically and socially.

Today, there is a growing proportion of geriatric individuals in society. According to 2015 data from the World Health Organization, 900 million geriatric individuals live on earth. According to a population projection made by the WHO in 2018, the elderly population is estimated to reach around 2 billion people out of 900 million people by 2050. These data show that 22% of society will be made up of older individuals by 2050.

There were no studies that investigated the effects of different living environments thoroughly on geriatric individuals.The purpose of this research is to evaluate and compare cognitive functions, balance, musculoskeletal pain level, psychological state, participation level in activities of daily living, and quality of life of elderly people living at home and elderly people living in nursing homes in Turkey.

The Aim of This Study Is: To assess and compare of cognitive function, balance, quality of life, depression and daily living activities of geriatric individuals, living in home environment and nursing home

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to research,
* Being in the age range of 65-95,
* Individuals with no known health problems, caused inactivity.
* Adequate cognitive functions (Standardized Mini Mental Test score of 24 and above).
* Individuals who do not have musculoskeletal problems that prevent physical activity.
* Giving the informed consent.

Exclusion Criteria:

* Mental retardation
* Epileptic history
* Those with diseases that cause neurological, orthopedic, and musculoskeletal problems.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Geriatric individuals, either living in home environment or a nursing home in Istanbul.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Cognitive performance evaluation | 10 minutes after obtaining socio-demographic information (It was done between the 10th and 25th minutes of the assessment)
  Standardized Mini Mental Test (SMMT) was used. It is used for the quantitative evaluation of cognitive performance within the standard neuropsychiatric examination methods. The test is a short, useful, and a standardized method that can be used globally to determine the cognitive level. It is evaluated in 11 items and under 5 main titles and over a total of 30 points. Low score refers to severe cognitive impairment.
Pain severity assessment | 25 minutes after obtaining socio-demographic information (It was done between the 25th and 30th minutes of the assessment)
  Visual Analogue Scale (VAS) that is an easy, reproducible, minimal tool-requiring, and understandable measurement tool for the assessment of pain intensity was used. This scale consists of a horizontal, straight line. There is a value of 0 at the beginning of the line and 10 at the end.
Balance assessment | 30 minutes after obtaining socio-demographic information. After the visual analogue scale evaluation, the geriatric individuals were rested for 5 minutes (It was done between the 35th and 50th minutes of the assessment).
  Berg Balance Scale (BDI) was used to measure balance performance in geriatric individuals. It is often used in clinical trials to assess postural control and predict the risk of falls. The test is made difficult by reducing the ground support. This test consists of 14 items and each section is rated between 0 (bad) and 4 (best). The high score indicates the best balance. 0-20 indicates high risk, 21-40 indicates moderate risk and 41-64 indicates low risk.
Evaluation of Depression score | 50 minutes after obtaining socio-demographic information (It was done between the 50th and 60th minutes of the assessment).
  Geriatric Depression Scale (GDS) was used. It consists of 30 self-report questions. In the scoring of the scale, 1 point is given to each answer that suggests depression, and 0 is given for the other answers, and the final score is considered as the depression score. A cut off value of 0-10 was defined as the absence of depression, 11-13 as "probable depression," and 14 and above as "definite depression."
Activities of daily living | 60 minutes after obtaining socio-demographic information. After the geriatric depression scale evaluation, the geriatric individuals were rested for 5 minutes. (It was done between the 65th and 70th minutes of the assessment).
  Barthel Index (BI) was used. The Barthel index consists of 10 main items. The items measure feeding, transferring from bed to wheelchair and to and from a toilet, grooming, bathing, walking on a level surface (or propelling a wheelchair if unable to walk), going up and down the stairs, dressing and undressing, controlling bladder and controlling bowel. The total score is between 0 and 100 and scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, 91-99 indicates "slight" dependency and 100 indicate "total" independency.
Assessment of Quality of life | It was completed after 70 minutes obtaining socio-demographic information.
  Short Form 36 (SF-36) was used. It is a scale that has a generic scale feature and provides extensive measurement. It consists of 36 questions under 8 subheadings. Low scores indicate deterioration in the quality of life.

SECONDARY OUTCOMES:
Body mass index | After the permission of patients, it was calculated, in the first 10 minutes of assessment.
  Body mass index (BMI) is an inexpensive and easy screening method for weight category. It was calculated with person's weight in kilograms divided by the square of height in meters.
Using of walking aids | After the permission of patients, it was calculated, in the first 10 minutes of assessment.
  Whether the participant used a walking aid or not was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yildiz Ozer, PT, PhD, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)